CLINICAL TRIAL: NCT06429735
Title: PRIME: An Early Feasibility Study of a Precise Robotically Implanted Brain-Computer Interface for the Control of External Devices
Brief Title: Precise Robotically IMplanted Brain-Computer InterfacE
Acronym: PRIME
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuralink Corp (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: N1-EFS-001
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Tetraplegia/Tetraparesis; Quadriplegia; Cervical Spinal Cord Injury; Amyotrophic Lateral Sclerosis; Quadriplegia/Tetraplegia; Tetraplegic; Paralysis
Keywords: spinal cord injury; SCI; BCI; brain computer interface; ALS; quadriplegia; tetraplegic; paralysis
MeSH Terms: conditions — Quadriplegia; Amyotrophic Lateral Sclerosis; Paralysis; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Neuralink N1 Implant and R1 Robot (Experimental): Implantation of the N1 Implant by the R1 Robot.
  Interventions: Device: N1 Implant; Device: R1 Robot

INTERVENTIONS:
Device: N1 Implant — The N1 Implant is a type of implantable brain-computer interface
  Other Names: Neuralink N1 Implant, N1, Telepathy, Link
Device: R1 Robot — The R1 Robot is a robotic electrode thread inserter that implants the N1 Implant.
  Other Names: R1, Neuralink R1 Robot

SUMMARY:
The PRIME Study is a first-in-human early feasibility study to evaluate the initial clinical safety and device functionality of the Neuralink N1 Implant and R1 Robot device designs in participants with tetraparesis or tetraplegia. The N1 Implant is a skull-mounted, wireless, rechargeable implant connected to electrode threads that are implanted in the brain by the R1 Robot, a robotic electrode thread inserter.

ELIGIBILITY:
Inclusion Criteria:

* Severe quadriplegia (tetraplegia) due to spinal cord injury or amyotrophic lateral sclerosis (ALS) for at least 1 year without improvement, where quadriplegia is defined as having very limited or no hand, wrist, and arm movement and all levels below
* Life expectancy ≥ 12 months.
* Ability to communicate in English
* Presence of a stable caregiver

Exclusion Criteria

* Moderate to high risk for serious perioperative adverse events
* Active implanted devices
* Morbid obesity (Body Mass Index > 40)
* History of poorly controlled seizures or epilepsy
* History of poorly controlled diabetes
* Requires magnetic resonance imaging (MRI) for any ongoing medical conditions
* Acquired or hereditary immunosuppression
* Use of smoking tobacco or other tobacco products
* Psychiatric or psychological disorder
* Brain MRI demonstrating hemorrhage, tumor, distorted or adverse anatomy.
* Any condition which, in the opinion of the Investigator, would compromise your ability to safely participate in the study or undergo the implantation procedure

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Device-Related Adverse Events (AE) | 12 months post-implant
Procedure-Related Adverse Events (AE) | 12 months post-implant

SECONDARY OUTCOMES:
Device-Related Adverse Events (AE) | Up to 72 months post-implant
Procedure-Related Adverse Events (AE) | Up to 72 months post-implant

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Ponce, MD, Principal Investigator — Barrow Neurological Institute; Jonathan Jagid, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - Barrow Neurological Institute, Phoenix, Arizona
  - University of Miami, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: https://neuralink.com/ — https://neuralink.com/